CLINICAL TRIAL: NCT05194319
Title: Determining the Effect of Upper Extremity Functional Skills on Quality of Life and Participation in Children With Diparetic Cerebral Palsy
Brief Title: Effect of Upper Extremity Functional Skills on Quality of Life and Participation of the Children With Cerebral Palsy
Acronym: CP
Status: Completed | Type: Observational
Sponsor: Sanko University (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Hatice Adiguzel, PT, Assistant Proffessor, Sanko University
Other Study IDs: SANKOO
Record Dates: First submitted 2022-01-03; First posted 2022-01-18 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Cerebral Palsy; Diplegia; Upper Extremity Dysfunction; Quality of Life; Participation, Patient
Keywords: Upper Extremity Functions; Diparetic Cerebral Palsy; Quality of Life; Participation
MeSH Terms: conditions — Cerebral Palsy; Patient Participation | interventions — Quality of Life

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1/Children with diparetic cerebral palsy: Children with diparetic cerebral palsy
  Interventions: Other: All assessments of children (Demographic information, upper extremity skills, quality of life and participation levels)
- 2/Healty control: Children with healty peer ages of cerebral palsy children.
  Interventions: Other: All assessments of children (Demographic information, upper extremity skills, quality of life and participation levels)

INTERVENTIONS:
Other: All assessments of children (Demographic information, upper extremity skills, quality of life and participation levels) — The researcher will fill out the personal information form containing the descriptive characteristics of the parents and children. GMFCS to assess children's functional levels, Manual Ability Classification System (MACS) to assess hand skills, Modified Ashworth Scale for upper extremity muscle spasticity, for upper extremity functional skills; Jebson Taylor Test, Abilhand Kids scale, for Quality of Life; The Quality of Life Scale for Children (PedsQL), PODCI criterion for participation levels will be administered by a physiotherapist who has 2 years of experience in the profession and works in the field of pediatric rehabilitation. The Jebson Taylor test and spasticity classification will be applied directly to the child by the physiotherapist, but other scales will be filled in by the parents under the supervision of the physiotherapist. .

SUMMARY:
Cerebral palsy (CP) is a movement and posture disorder accompanied by sensory, perception, cognition, communication and behavioral disorders that cause activity limitations by causing various non-progressive disorders of the fetal or infant brain. Spastic CP, according to the affected area in the body; It is classified as hemiparetic, diparetic and is observed most frequently. Diparetic CP, on the other hand, is characterized by significant spasticity in the pelvis and lower extremities, mild hypertonus or spasticity in the upper extremities, and incoordination, mostly involving the lower extremities and some upper extremities.Although lower extremity involvement is observed in different degrees in children with diparetic CP, studies showing how upper extremity and hand functions are affected are insufficient.The aim of this study is to compare the effect of upper extremity functional skills on quality of life and participation levels in children with diparetic CP with their healthy peers.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a movement and posture disorder accompanied by sensory, perception, cognition, communication and behavioral disorders that cause activity limitations by causing various non-progressive disorders of the fetal or infant brain. Spastic CP, according to the affected area in the body; It is classified as hemiparetic, diparetic and is observed most frequently. Diparetic CP, on the other hand, is characterized by significant spasticity in the pelvis and lower extremities, mild hypertonus or spasticity in the upper extremities, and incoordination, mostly involving the lower extremities and some upper extremities. Although lower extremity involvement is observed in different degrees in children with diparetic CP, studies showing how upper extremity and hand functions are affected are insufficient.Upper extremity functions are one of the most important factors that ensure participation in daily life for these children. Hands play a key role in the execution of activities of daily living (ADL), as well as being among the most important components affecting upper extremity functionality.Children with spastic type CP experience limitations in mobility due to the decrease in selective motor control, and as a result, they may experience losses in social life and limitations in participation in their ADLs. These children have various functional disabilities such as various gait disorders, lower extremity contractures and strength losses, trunk and postural control deficiencies, mobility problems, vision problems, behavioral and sensory problems, upper extremity strength and skill losses that affect school success. This situation causes them to encounter difficulties in taking an active role in life.

Quality of life is a concept that shows the personal reactions to diseases that affect the level of personal satisfaction and to the physical, mental and social effects of daily life.Evaluation of quality of life in children with CP mostly includes physical symptoms, activity limitation, emotional stress, communication problems between child and family, limitation of school life, and determination of difficulties in the treatment of the disease. Decreased functional independence in children with CP compared to their healthy peers with typical development. Difficulties in activities of daily living, accompanying cognitive and sensory problems negatively affect quality of life.However, studies examining the relationship between upper extremity functional skills, quality of life and participation level in children with diparetic CP are insufficient in the literature.The aim of this study is to compare the effect of upper extremity functional skills on quality of life and participation levels in children with diparetic CP with their healthy peers.

ELIGIBILITY:
Inclusion Criteria:

* To be between the ages of 6-15,
* Having the verbal communication ability to understand the evaluation materials and being willing to participate in the study (Written consent form will be obtained from the families), Being at the level of 1-3 when evaluated according to the GMFCS (Gross Motor Function Classification System),
* ≤ 2 in upper extremity muscles according to Modified Ashworth Scale (MASH)
* Being at 1-2 levels when evaluated according to MACS (Manual Ability Classification System),
* Absence of any contracture in the upper extremity
* Not having had any upper extremity surgery or Botulinum Toxin (Btx) in the last 6 months

Exclusion Criteria:

* Severe cognitive dysfunction or inability to communicate cognitively,
* Having a diagnosis of mental disability,
* Mothers are illiterate

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: diparetic cerebral palsy children between 6-15 years old and their healty peer aged children
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
The Jebsen-Taylor Hand Function Test (JTHFT) | first day of assessment
  JTHFT evaulates the upper extremity functional skills.Jebsen Taylor Hand Function Test (JTHFT) is a test used between the ages of 6 and 90, administered between 15 and 45 minutes, consisting of 7 items, using a scaled board to ensure the standard arrangement of the objects used and a stopwatch to measure the time when the activities are done. Test materials; dessert spoon, bean grain, soda bottle cap, coin, checker stone, light and heavy tin can, pen and writing materials. Before the application, the child is shown how to make the items in the test. Explaining that the test is done against time is necessary for the motivation of the child. The child starts the activity with the start command and the stopwatch is stopped as soon as he/she finishes that activity. If he fails the activity, that part of the test is not continued. Increasing test completion time indicates worse hand function.
ABILHAND-Kids | first day of assessment
  ABILHAND-Kids evaulates the assessment of upper extremity functional skills. Abilhand Kids is a 21-item functional test, mostly consisting of bimanual activities, answered by parents, assessing how children with CP aged 6-15 do their daily activities. With this questionnaire, parents evaluate the difficulty level of their children while doing an activity on a three-level scale as impossible, difficult and easy. Activities not done in the last 3 months are not scored within the scope of this survey and are considered as incomplete answers. Scores are '0 = Impossible', '1 = Difficult' and '2 = Easy'. A maximum of 42 points can be obtained in the test.
Pediatric Quality of Life Inventory (PedsQL) | first day of assesment
  Pediatric Quality of Life Inventory (PedsQL) evaulates the quality of life of the children with cp. It consists of 23 items. It questions physical health, emotional functioning, social functionality and school functionality. Scoring is done in 3 areas. First, the total score of the scale, secondly the total score of physical health, and thirdly, the total score of psychosocial health, which consists of calculating the item scores evaluating emotional, social and school functionality, is calculated.Items are scored between 0-100. A score of 100 is scored if the answer is marked as never, 75 if it is marked as rarely, 50 if it is marked as sometimes, 25 if it is marked as often, and 0 if it is marked as almost always. As a result, the higher the total PedsQL score, the better the health-related quality of life is perceived.
Pediatric Outcome Data Collection İnstrument (PODCI) | first day of assesment
  PODCI evaulates the participation level of the children with cp. The PODCI scale is used to determine the functional health status, physical functionality and participation level of children with CP. In addition to the evaluation of emotional and physical functions, it also reveals the expectations of families from the treatment applied to their children. The criterion can be applied to individuals aged 2-18 years. PODCI has 2 parent forms (child and adolescent) and adolescent form consisting of the same questions. The test is a Likert-type scale and consists of 6 sections: Upper Extremity Functions-UEF, Physical Function and Sports-FFS, Transfer and Basic Mobility-TM, Pain-RA, Happiness/Satisfaction-MM, and global function-GFR. Each of the sections is calculated from 0-100.

SECONDARY OUTCOMES:
demographic information | first day of assessment
  demographic information of the children and parents
Manual Ability Classification System (MACS) | first day of assessment
  Manual Skills Classification System of the children with cp. MACS; It is a five-level system developed by Elliason et al. in 2003 to classify the ability to handle objects during daily activities in children with CP aged 4-18 years. The determination of the levels is based on the child's ability to hold objects to himself and the need for assistance and adaptation in performing manual activities in daily life. A higher score indicates worse hand function.
GMFCS (Gross Motor Function Classification System) | first day of assessment
  Gross Motor Function Classification System of the children with cp. The main criterion while defining the five-level classification system is that the differences between the levels are meaningful in daily life. The differences are based on functional limitations, the need for hand-held mobility aids (walker, crutches, or canes) or wheeled mobility devices, and less so on the quality of movement. Higher level indicates worse functional level.
Modified Ashworth Scale | first day of assessment
  Classification of spasticity of upper extremity muscles of children with CP.This scale was developed to measure muscle tone. The resistance to passive movement is evaluated. It is scored between 0-4.
  0 No tone increase.
  1 There is a slight increase in muscle tone. When the affected part is flexed or extended, minimal resistance is felt at the end of the movement or there is a catch-and-release sensation.
  1+ Pulling sensation during movement, resistance felt in less than half of joint movement.
  2 Resistance is felt during most of the joint movement, but the affected part is easily moved.
  Passive movement is difficult throughout the 3 ROM. 4 The affected part is rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: Nevin Ergun, Proffessor, Study Director — Sanko University; Hatice Adıgüzel, PhD, Study Chair — Kahramanmaras Sutcu Imam University; merve Kafa, PT, Principal Investigator — Sanko University
Locations (1):
- Outpatient Rehabilitation Center, Gaziantep, Sahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No